CLINICAL TRIAL: NCT04935567
Title: PRediction of Vagal Nerve Stimulation EfficaCy In Drug-reSistant Epilepsy: Prospective Study for Pre-implantation Prediction
Brief Title: PRediction of Vagal Nerve Stimulation EfficaCy In Drug-reSistant Epilepsy
Acronym: PRECISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Collaborators: St. Anne's University Hospital Brno, Czech Republic (Other); University Hospital, Motol (Other); Na Homolce Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRECISE-21
Record Dates: First submitted 2021-05-18; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Drug Resistant Epilepsy
Keywords: Drug-resistant epilepsy; Vagal nerve stimulation; Efficacy predictability; Responders; Non-responders; EEG
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Models, Statistical

STUDY DESIGN:
Intervention Model Description: PRECISE is a prospective multicentre study for prediction VNS efficacy based on pre-implantation EEG data. The patients with drug-resistant epilepsy will undergo standard VNS implantation based on a clinical decision. Before implantation, the scalp EEG, according to the study protocol, will be recorded. The EEG will be mathematically processed, and the patient´s predicted outcome in terms of predicted responder vs. predicted non-responders will be statistically determined. The stimulation parameters and AEDs therapy will be modified according to the best clinical practice. The real-life outcome will be determined by percent seizure reduction. Subsequently, the real-life and predicted outcome will be compared in terms of accuracy, sensitivity, and specificity. The main goal is to validate Pre-X-Stim in a real-life prospective study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Predicted responders (Experimental): Patients indicated VNS therapy as their standard for clinical care and are concerned about the prediction of VNS efficacy based on pre-implantation EEG, (≥50% seizure reduction).
  Interventions: Other: Statistical model for the prediction of VNS efficacy
- Predicted non-responders (Active Comparator): Patients indicated VNS therapy as their standard for clinical care and are concerned about the prediction of VNS efficacy based on pre-implantation EEG, (<50% seizure reduction).
  Interventions: Other: Statistical model for the prediction of VNS efficacy

INTERVENTIONS:
Other: Statistical model for the prediction of VNS efficacy — statistical model for the prediction of VNS efficacy based on a mathematical and statistical analysis of scalp EEG data
  Other Names: the verification of the real-life validity of the statistic classifier for prediction of VNS response based on pre-implantation EEG

SUMMARY:
Vagal nerve stimulation (VNS) can be indicated in patients with drug-resistant epilepsy who are not eligible for resective epilepsy surgery with responders rates about 50% (≥50% seizure reduction). At the moment, there is not a widely-accepted possibility to predict VNS efficacy in a given patient based on pre-implantation data, which can lead to unnecessary surgery and improper allocation of financial resources. The principal aim of PRECISE (PRediction of vagal nerve stimulation EfficaCcy In drug-reSistant Epilepsy) study is to verify the predictability of VNS efficacy by analysis of pre-implantation routine EEG. The PRECISE relies on the results of our previous work, which developed a statistical classifier for VNS response (responders vs. non-responders) based on differences in EEG power spectra dynamics (Pre-X-Stim). PRECISE is designed as a prospective multicentre study in which patients indicated to VNS therapy will be recruited. Patients will be classified as predicted responders vs. predicted non-responders using pre-implantation EEG analyses. After the first and the second year of the study, the real-life outcome (responder vs. non-responder) will be determined. The real-life outcome and predicted outcome will be compared in terms of accuracy, specificity, and sensitivity. In the meantime, the patients will be managed according to the best clinical practice to obtain the best therapeutical response.

DETAILED DESCRIPTION:
The patients will be recruited within cooperating epilepsy centres. The recruitment limited to cooperating centres will ensure the correct indication for VNS therapy and the adjustment of VNS parameters according to the best medical practice, which are not part of the study protocol itself, but are crucial for the study results.

The VNS will be indicated in a given patient based on a clinical decision as a standard of patient´s therapy (i.e., the indication of VNS is not a part of the proposed project). The patient will be informed about the study on a pre-implantation visit or by a phone call, during which initial eligibility for the study will be determined, and study protocol and design will be explained by research staff.

G. Assessment 0 - pre-implantation assessment Assessment 0 includes screening for eligibility criteria and obtaining baseline data on subjects participating in the study. After the signature of informed consent, the patient will be given a unique code by which all data will be labelled. The demographic information, health history, including psychiatric disease and type of epilepsy, concomitant medication (AEDs and other drugs), and seizure frequency will be collected. The seizure frequency will be analysed based on the patient diary. Standard EEG will be recorded according to the protocol described below.

Protocol for EEG recording The EEG will be recorded on the EEG recording system with a sampling frequency of 250 Hz or higher, with electrodes placed on the scalp according to 10-20 system (electrodes names as follows: Fp1, Fp2, F7, F3, Fz, F4, F8, T3, C3, Cz, C4, T4, T5, P3, Pz, P4, T6, O1, and O2). Different electrodes names are allowed, but their position must correspond with the position of previously defined electrodes. Additional electrodes are also allowed, but will not be evaluated within the study. EEGs with lower numbers or different positions of electrodes are not allowed.

The EEG is recorded in a supine position with eyes closed except for periods with eyes opening. The recorded EEG will have a duration of 20 minutes or more and must contain defined segments in the following order (Figure 1):

Segment 1 - Rest 1 - duration at least 2 min Segment 2 - Eyes opening/closing - duration at least 10 s Segment 3 - Rest 2 - duration at least 10 s; immediately after eye closure Segment 4 - Photic stimulation - stimulation frequencies: 5 Hz (10 s) - 10 Hz (10 s) - 15 Hz (10s) - 20 Hz (10 s) - 25 Hz (10 s) - 30 Hz (10 s) - 25 Hz (5 s) - 20 Hz (5 s) - 15 Hz (5 s) - 10 Hz (5 s) - 5 Hz (5 s); light intensity at least 0.7 Joule Segment 5 - Hyperventilation - duration at least 4 min (2 minutes hyperventilation by nose + 2 minutes hyperventilation by mouth) Segment 6 - Eyes opening/closing - duration at least 10 s Segment 7 - Rest 3 - duration at least 10 s, immediately after eye closure Segment 8 - Rest 4 - duration at least 2 minutes The recorded EEG will be anonymized and labelled by a unique code previously attributed to a patient. In the next step, the EEG will be sent for mathematical/statistical processing. Based on this processing, the patients´ predicted response to VNS will be determined in terms of predicted responders (seizure reduction ≥ 50%) vs. predicted non-responders (seizure reduction < 50%). Neither the patient nor the physician will be informed about the classification results.

Follow-up assessments - Assessments 1, 2 Two assessments are designed in patients´ follow-up: Assessment 1 - 1 year after stimulation initialization and Assessment 2 - 2 years after stimulation initialization.

Assessment 1, 2 The patients will be evaluated 1 and 2 years after stimulation initialization. The patient will be asked about changes in health history, including psychiatric disease, concomitant medication (AEDs and other drugs), VNS parameters setting, and seizure frequency. The seizure frequency will be collected by reviewing patients 'diary. The reported seizure frequency will be compared with pre-implantation seizure frequency, and real-life response will be calculated in terms of real-life responders (seizure reduction ≥ 50%) or real-life non-responder (seizure reduction < 50%). If the patient does not tolerate at least the minimal VNS setting (0.75 mA) because of serious adverse events, he/she will be excluded from further analysis (the patient´s data will be reported separately).

The information collected in Assessment 1 and 2, including real-life response to VNS, will be labelled by the patient´s unique code and will be sent to the coordinating centre, where it will be compared with the patient´s predicted response.

At the end of Assessment 2, the patient will be asked if he/she is interested in the predicted response to VNS. If yes, the study physician will contact the coordinating centre, where the predicted response for a given patient will be conveyed. The patient will be informed about the predicted response by a phone call or during a regular visit (not a part of the study protocol, described below).

The study is concerned with the verification of the real-life validity of our statistic classifier for the prediction of VNS response based on pre-implantation EEG. The patients based on the pre-implantation EEG will be classified based on their predicted response as predicted responders (≥50% seizure reduction) vs. predicted non-responders (<50% seizure reduction). In Assessment 1 a 2, respectively, the patients´ real-life response will be determined: real-life responders (≥50% seizure reduction) vs. real-life non-responder (< 50% seizure-reduction). The predicted and real-life responses will be statistically compared in terms of accuracy, sensitivity, and specificity.

The individual patients´ groups (predicted responders vs. predicted non-responders, real-life responders vs. real-life non-responders) will be compared based on their demographic data, health history, AEDs, and VNS parameter. A suitable statistical test will be chosen concerning the data´s characteristics (Pearson´s Chi-squared test for categorical variables, Wilcoxon-Mann-Whitney test for continuous variables).

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant epilepsy indicated to VNS based on clinical decision.
* Drug-resistant epilepsy is defined as a failure of adequate trials of two tolerated, appropriately chosen, and used antiepileptic drug schedules (whether as monotherapy or in combination) to achieve sustained seizure freedom (Kwan et al., 2010).
* Age ≥ 18 years
* Availability to record 20 minutes of EEG with photic stimulation, hyperventilation, and eye-opening/closing according to the pre-defined protocol.
* Availability of seizure diaries at least three months before VNS implantation OR reliable information about seizure frequency at least three months before VNS implantation
* The ability of a patient/family member/caregiver to record seizures precisely into seizure diaries OR the ability of a patient/family member/caregiver to report seizures precisely different ways.
* In cases with very high seizure frequency (several seizures per day), it is acceptable to report only the days without any seizures.

Exclusion Criteria:

* The indication and planning of resection brain surgery as a treatment option for drug-resistant epilepsy. If a patient clearly demonstrates his refusal of resection surgery, he/she can be included in the study.
* The presence of psychogenic non-epileptic seizures which cannot be reliably distinguished from epileptic seizures by a patient/family member/caregiver.
* The presence of other condition which can resemble epileptic seizures which cannot be reliably distinguished from epileptic seizures by a patient/family member/caregiver.
* Metabolic condition or other diseases, in which the increase of seizure frequency is expectable.
* The inability of a patient to take regular visits which are required for VNS parameters settings or the study
* Life expectancy shorter than two years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of statistic model for prediction of response to VNS therapy | 2 years
  Accuracy of statistic model for prediction of response to VNS therapy in terms of responders and non-responders in drug-resistant epilepsy

SECONDARY OUTCOMES:
The quantification of differences in EEG power spectra | 2 years
  The quantification of differences in EEG power spectra (Relative Mean Power, %) between real-life responders and real-life non-responders to VNS therapy in drug-resistant epilepsy
Prediction of patients' response to VNS therapy | 2 years
  Prediction of patients' response to VNS therapy in terms of responders (≥ 50% seizure reduction from baseline) and non-responders (<50% seizure reduction from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Brazdil, Prof., Principal Investigator — University Hospital st. Anne´s Brno
Locations (1):
- University Hospital St. Anne´s Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dolezalova I, Koritakova E, Souckova L, Chrastina J, Chladek J, Stepanova R, Brazdil M. Prediction of Vagal Nerve Stimulation Efficacy in Drug-Resistant Epilepsy (PRECISE): Prospective Study for Pre-implantation Prediction/Study Design. Front Neurol. 2022 Mar 21;13:839163. doi: 10.3389/fneur.2022.839163. eCollection 2022. PMID 35386419